CLINICAL TRIAL: NCT01186549
Title: Title: The Effect of Combined Ephedrine and Lidocaine Pretreatment on Pain Due to Propofol Injection in Patients Undergoing Elective Surgery Under General Anaesthesia
Brief Title: The Effect of Combined Ephedrine and Lidocaine Pretreatment on Pain and Hemodynamic Changes Due to Propofol Injection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Qazvine University Of Medical Sciences, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12610000610033; ACTRN12610000610033
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Pain Due to Propofol Injection; Hemodynamic Changes Due to Propofol Injection
Keywords: propofol; ephedrine; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ephedrine 30 microgram/kg (Active Comparator): Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Interventions: Drug: Ephedrine 30microgram/kg
- ephedrine 70 microgram/kg (Active Comparator): Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Interventions: Drug: ephedrine 70 microgram/kg
- lidocaine0.5mg/kg -ephedrine30 micrograms/kg (Active Comparator): Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Interventions: Drug: lidocaine0.5mg/kg -ephedrine30 micrograms/kg
- lidocaine 0.5mg/kg (Active Comparator): Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Interventions: Drug: lidocaine 0.5mg/kg
- normal saline 2ml (Placebo Comparator): Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Interventions: Drug: normal saline 2ml

INTERVENTIONS:
Drug: Ephedrine 30microgram/kg — Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Arms: ephedrine 30 microgram/kg
Drug: lidocaine0.5mg/kg -ephedrine30 micrograms/kg — Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Arms: lidocaine0.5mg/kg -ephedrine30 micrograms/kg
Drug: ephedrine 70 microgram/kg — Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Arms: ephedrine 70 microgram/kg
Drug: lidocaine 0.5mg/kg — Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Arms: lidocaine 0.5mg/kg
Drug: normal saline 2ml — Patients were randomly allocated to one of 5
  groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30micrograms/kg (E30)ephedrine 70micrograms/kg(E70),lidocaine0.5mg/kg -ephedrine30 micrograms/kg(LE) or 2ml saline (S)intravenously.participants in each group receive a single dose of the intervention treatment only.After one minute propofol 2 mg/kg into a dorsal hand vein was injected
  Arms: normal saline 2ml

SUMMARY:
Objectives: Injection pain and hypotension are two main adverse effects of propofol which distresses patient. The aim of this prospective double blind study was to compare the effect of ephedrine -lidocaine combination with lidocaine and ephedrine on injection pain and hemodynamic changes due to propofol induction.

Methods: 165 adult patients, aged 20 to 60 yr, Patients were randomly allocated to one of 5 groups (33 patients per group): lidocaine 0.5 mg/kg(L) ,ephedrine 30microgram/kg (E30), ephedrine 70 microgram/kg(E70), lidocaine 0.5mg/kg -ephedrine 30 microgram/kg(LE) or 2ml saline (S) intravenously. After one minute propofol 2 mg/kg into a dorsal hand vein was injected. Face pain scale and verbal rating scale, arterial blood pressure and heart rate were recorded before induction, just before intubation, and one minute after intubation

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists(ASA)physical statusIandII

Exclusion Criteria:

* patients with difficulty in communication
* history of allergic, neurologic or cardiovascular disease
* patients who had received an analgesic medication within 24 hr before surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
pain during propofol injection is assessed by face pain scale(FPS) and verbal rating scale(VRS) | during the injection period of propofol(One minute after the administration of the test solution) before loss of consciousness

SECONDARY OUTCOMES:
mean arterial blood pressure | before the administration of the test solution , just before intubation(three minutes after atracurium injection), and one minute after intubation
  mean arterial blood pressure is assessed by nonivasive automatic blood pressure measurement
heart rate | before the administration of the test solution, just before intubation(three minutes after atracurium injection) , and one minute after intubation
  is assessed by echocardiogram monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin university of medical science, Qazvin, Qazvin Province, Iran